CLINICAL TRIAL: NCT00303407
Title: Prophylaxis of Venous Thrombo-Embolism in Cancer Patients Under Palliative Care
Status: Terminated | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Other Study IDs: SPOT 99/54
Record Dates: First submitted 2006-03-15; First posted 2006-03-16 (Estimated); Last update posted 2006-03-16 (Estimated); Status verified 2005-12

CONDITIONS: Cancer; Venous Thromboembolism
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism | interventions — Nadroparin

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: nadroparin

SUMMARY:
To determine the efficacy and to measure the complications of prophylactic anticoagulation using low-molecular weight heparin in adult cancer patients under palliative care

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients in palliative care
* Patients fully informed about their condition
* Signed informed consent
* No exclusion criteria

Exclusion Criteria:

* Absence of advanced cancer
* Cancer previously cured
* Venous thromboembolism diagnosed within 6 months prior to inclusion
* Absence of discerning capacity
* Active anti-thrombotic treatment with heparins or coumarines
* Thrombocytopenia <50G/l
* PTT >45sec
* TP<35%
* Active bleeding
* Renal failure <20ml/min
* Past history of heparin-induced thrombocytopenia

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-01; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Weber, MD, Principal Investigator — Center of Continuous Care, chemin de la Savonnière 11, CH-1245 Collonge-Bellerive
Locations (1):
- Center of Continuous Care, chemin de la Savonnière, Collonge-Bellerive (Geneva), Canton of Geneva, Switzerland

REFERENCES:
- [Background] Prandoni P. Antithrombotic strategies in patients with cancer. Thromb Haemost. 1997 Jul;78(1):141-4. PMID 9198144